CLINICAL TRIAL: NCT00000785
Title: A Registry of Tuberculosis Cases in the CPCRA
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 017; 11568 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Tuberculosis; Mycobacterium tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome; Drug Resistance, Microbial
MeSH Terms: conditions — HIV Infections; Tuberculosis; AIDS-Related Opportunistic Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Any sample that can be used to test for M.tuberculosis

GROUPS / COHORTS (1):
- A: All eligible CPCRA subjects

SUMMARY:
PRIMARY: To estimate the proportion of tuberculosis patients in the CPCRA who have drug-resistant tuberculosis (TB) and to describe the patterns of drug resistance.

SECONDARY: To compare drug resistance data on the Mycobacterium tuberculosis isolates of HIV-infected patients to those of HIV-uninfected patients who are being followed in the CPCRA. To assess the relationship of resistance data with geographic, demographic, and HIV and TB risk factor information.

Geographic areas and demographic subgroups affected by the TB epidemic appear to be congruent and associated with the concurrent HIV epidemic. The total number of CPCRA patients who will develop, or who have experienced, confirmed TB is unknown. It is critical to determine the depth and breadth of the current problem of drug-resistant TB.

DETAILED DESCRIPTION:
Geographic areas and demographic subgroups affected by the TB epidemic appear to be congruent and associated with the concurrent HIV epidemic. The total number of CPCRA patients who will develop, or who have experienced, confirmed TB is unknown. It is critical to determine the depth and breadth of the current problem of drug-resistant TB.

For both retrospective and prospective components of the study, demographic, geographic, HIV and TB risk factor information will be collected on CPCRA patients with confirmed pulmonary or extrapulmonary TB. Mycobacterial culture results will be recorded. Retrospective data will be collected on CPCRA patients with confirmed tuberculosis who have been diagnosed since January 1992 until the time of site registration. Prospective data will be collected on CPCRA patients with confirmed tuberculosis diagnosed during the period of 1 to 2 years following site registration.

ELIGIBILITY:
Patients must meet the following criteria:

* CPCRA patients with confirmed pulmonary or extrapulmonary TB. Confirmed clinical TB requires a positive culture for Mycobacterium tuberculosis.

NOTE:

* There is no requirement that patients have HIV infection.

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All eligible CPCRA subjects
Sampling Method: Non-Probability Sample
Enrollment: 1509 (Actual)
Dates: Start 1992-08; Primary Completion 1994-06 (Actual); Study Completion 1994-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred Gordin, Study Chair
Locations (13):
- United States (13):
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Gordin FM, Nelson ET, Matts JP, Cohn DL, Ernst J, Benator D, Besch CL, Crane LR, Sampson JH, Bragg PS, El-Sadr W. The impact of human immunodeficiency virus infection on drug-resistant tuberculosis. Am J Respir Crit Care Med. 1996 Nov;154(5):1478-83. doi: 10.1164/ajrccm.154.5.8912768.